CLINICAL TRIAL: NCT07090733
Title: The Effect of Ultrasound Guided Interscalene, Suprascapular and Anterior Glenoid Nerve Blocks on Diaphragmatic Excursion and Analgesia Following Arthroscopic Shoulder Surgery: A Prospective Randomized Controlled Study
Brief Title: Ultrasound Guided Interscalene, Suprascapular and Anterior Glenoid Nerve Blocks on Diaphragmatic Excursion and Analgesia Following Arthroscopic Shoulder Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Fatma Elsamahy, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36265MD/12/24
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Interscalene Block; Suprascapular Nerve Block; Anterior Glenoid Nerve Block; Diaphragmatic Excursion; Analgesia; Arthroscopic Shoulder Surgery
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Active Comparator): Patients will receive general anesthesia, plus an ultrasound-guided Interscalene brachial plexus block (ISB) with the injection of 15 mL of 0.25% bupivacaine.
  Patients will receive general anesthesia plus an ultrasound-guided suprascapular nerve block (SSNB)
  Interventions: Other: Interscalene brachial plexus block
- Group II (Experimental): Patients will receive general anesthesia plus an ultrasound-guided suprascapular nerve block (SSNB) with injection of 15 ml of 0.25% bupivacaine.
  Interventions: Other: Suprascapular nerve block
- Group III (Experimental): Patients will receive general anesthesia plus an ultrasound-guided anterior glenoid block with injection of 15 ml of 0.25% bupivacaine.
  Interventions: Other: Anterior glenoid block
- Group IV (Experimental): Patients will receive general anesthesia, along with a total volume of 30 mL of bupivacaine 0.25%, divided into 15 mL of Bupivacaine 0.25% for ultrasound-guided SSNB and 15 mL of Bupivacaine 0.25% for ultrasound-guided anterior glenoid block.
  Interventions: Other: Suprascapular nerve block + Anterior glenoid block

INTERVENTIONS:
Other: Interscalene brachial plexus block — Patients will receive general anesthesia, plus an ultrasound-guided interscalene brachial plexus block (ISB) with the injection of 15 mL of 0.25% bupivacaine.
  Other Names: 15 ml of 0.25% bupivacaine
  Arms: Group I
Other: Suprascapular nerve block — Patients will receive general anesthesia plus an ultrasound-guided suprascapular nerve block (SSNB) with injection of 15 ml of 0.25% bupivacaine.
  Other Names: 15 ml of 0.25% bupivacaine
  Arms: Group II
Other: Anterior glenoid block — Patients will receive general anesthesia plus an ultrasound-guided anterior glenoid block with injection of 15 ml of 0.25% bupivacaine.
  Other Names: 15 ml of 0.25% bupivacaine
  Arms: Group III
Other: Suprascapular nerve block + Anterior glenoid block — Patients will receive general anesthesia, along with a total volume of 30 mL of 0.25% bupivacaine, divided into 15 mL for ultrasound-guided SSNB and 15 mL for ultrasound-guided anterior glenoid block.
  Other Names: 30 mL of 0.25% bupivacaine
  Arms: Group IV

SUMMARY:
This study aims to evaluate the diaphragmatic movement and postoperative analgesia following anterior glenoid, suprascapular, and interscalene nerve blocks in patients undergoing elective arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
Arthroscopic shoulder surgery is a key approach for diagnosing and treating many shoulder disorders. Nevertheless, 30-70% of patients often experience moderate to severe pain, especially at 48 h after the operation, which affects rapid recovery.

The interscalene brachial plexus block (ISB) remains the gold standard for providing analgesia after shoulder surgery. Suprascapular nerve block (SSNB) is the most commonly used regional nerve block. Seventy percent of the sensory nerve fibers of the shoulder joint are innervated by the suprascapular nerve (SSN), with the supraspinatus and infraspinatus being directly innervated by the SSN.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I or II.
* Scheduled for arthroscopic shoulder surgery.

Exclusion Criteria:

* Patient's refusal to participate.
* Patients with a history of allergy to local anesthetics.
* Patients with a history of chronic use of painkillers.
* Patients presented with mental dysfunction.
* Patients with coagulation disorders.
* Patients presented with skin or soft tissue infection at the proposed site of needle Insertion.
* Pregnant Patients.
* Patients with Chronic Obstructive Pulmonary Disease (COPD) or a Body Mass Index (BMI) of more than 40.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hemi-diaphragmatic paralysis | 24 hours postoperatively
  Incidence of hemi-diaphragmatic paralysis determined by ultrasound-guided assessment of diaphragmatic excursion. Diaphragmatic excursion will be measured before procedure (pre-block), 30 minutes after performing the block and post operative after complete recovery in post-anesthesia care unit (PACU).

SECONDARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numerical rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be recorded at T0, 30 min, 2, 4, 6, 12, 18, and 24 hours postoperatively.
Total analgesic consumption | 24 hours postoperatively
  All patients will receive Paracetamol 1 g/6 hours as a regular analgesia and Morphine 3mg if the numerical rating scale (NRS) > 3 as a rescue analgesia.
Degree of patient satisfaction | 24 hours postoperatively
  The degree of patient satisfaction will be assessed based on a questionnaire and graded on a 4-point scale (excellent/good/fair/poor)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.